CLINICAL TRIAL: NCT06674278
Title: Changes in Electrocardiographic (ECG) Ventricular Repolarization and Transthoracic Impedance Cardiography (ICG) Parameters in Patients with COVID-19 and After the Disease: Persistence and Prognostic Significance of These Changes
Status: Not yet recruiting | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jonas Jucevičius, Investigator, Assistant lecturer., Lithuanian University of Health Sciences
Other Study IDs: BE-2-40
Record Dates: First submitted 2024-10-15; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-05

CONDITIONS: Post COVID-19; Ventricular Repolarization; Arrhythmias; Impedance Cradiography
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with changes in ECG repolarization parameters and arrhythmias during acute COVID-19
- Patients without changes in ECG repolarization parameters and arrhythmias during acute COVID-19

SUMMARY:
The aim of this study is to determine the relationship between changes in resting electrocardiography (ECG) ventricular repolarization parameters, transthoracic impedance cardiography (ICG) parameters, and COVID-19, to assess the relationship between ECG changes after COVID-19 and heart rhythm disorders (arrhythmias), cardiovascular events (the onset and exacerbation of cardiovascular diseases), the persistence of changes two years after the illness, and to identify prognostic ventricular repolarization parameters in patients with and after COVID-19.

It is expected that the results obtained during the study will help predict long-term cardiovascular complications in these patients, aiming to prevent them by providing recommendations for the long-term monitoring of individuals who have recovered from COVID-19. Additionally, the investigators hope to propose a new ECG ventricular repolarization parameter that could be used in the future for prognostic assessment in patients with other diseases as well.

DETAILED DESCRIPTION:
Purpose:

To find the relation between changes in resting electrocardiography (ECG) ventricular repolarization parameters and the consequences of COVID-19. To assess these parameters connection with arrhythmias and overall cardiovascular events and transthoracic impedance cardiography (ICG) parameters, to evaluate the persistence of changes over a 2-year period after the illness, and to identify prognostic ventricular repolarization and ECG parameters in COVID-19 patients.

Goals of the study:

1. To identify the most common differences in ECG ventricular repolarization parameters among COVID-19 patients who experienced arrhythmias and/or other cardiovascular events within 2 years of hospital discharge, compared to those who did not have arrhythmias and/or other cardiovascular events.
2. To assess the persistence of changes in ECG ventricular repolarization parameters 2 years after hospital discharge.
3. To identify and determine the differences in ICG parameters among individuals who have recovered from COVID-19 2 years after their hospital discharge.
4. To find the most appropriate prognostic ECG criteria for monitoring recommendations for patients who have recovered from COVID-19.

Duration of the study: the study is estimated to take 3 years (from 2024 11 to 2027 09). Each enrolled participant participates in study for 2 days (a little more than 24 hours total): one hour is allocated for the examination (taking medical history, objective examination, ECG, echocardiography, placing the Holter monitoring device, and performing the ECG) and the following day for about 5 minutes when participant returns for the removal of the Holter monitoring device.

Methods. Study design: this is a prospective, nested case-control study.

Patients who had COVID-19 since January 1, 2022, and were treated in the LUHS Kaunas Hospital 2 years ago (beginning January 1, 2022), are invited to participate in the study if they consent to be enrolled, meet the selection criteria, and do not have any exclusion criteria. The enrollment will last until the required sample size is collected.

The following data is going to be collected: age, anthropometric data (height, weight), detailed history of COVID-19 (including previous illnesses, vaccination status), history of comorbidities (chronic cardiovascular diseases, particularly detailed history of arrhythmias and overall cardiovascular events over the last two years, including conduction disorders, also lung diseases, diabetes, kidney and urinary system diseases, hematological diseases, gastrointestinal diseases, connective tissue, joint, systemic diseases, infectious diseases), history of harmful habits, and history of medications used (including those taken during hospitalization).

Anamnestic and examination data will be assessed based on participants records, including ECG performed during hospitalization, imaging studies (chest X-ray), and laboratory tests. Information about medications prescribed during treatment will also be collected. Cardiovascular events, episodes of arrhythmias, and conduction disturbances over the last 2 years after COVID-19 will also be evaluated retrospectively.

An objective examination focusing on the cardiovascular system will be performed (blood pressure, heart rate, heart auscultation findings).

Participants will undergo a resting 12-lead ECG. The following parameters will be assessed- left/right ventricular hypertrophy, arrhythmias (sinus, supraventricular, and ventricular types), conduction abnormalities, ischemia/infarction signs, QRS duration. Parameters of ventricular repolarization such as QT, QTc, Tpe, Tpec, Tpe/QT, Tpec/QTc, and the QRS-T angle will be evaluated.

Transthoracic echocardiography will be performed to assess signs of ventricular hypertrophy, systolic and diastolic left ventricular function, right ventricular function, atrial abnormalities, signs of pulmonary hypertension and heart valve pathology.

A transthoracic impedance cardiography (ICG) will be performed focusing on the thoracic fluid capacity, thoracic fluid volume index, systemic vascular resistance, and systemic vascular resistance index.

24-hour ECG Holter monitoring will be performed to evaluate arrhythmias (sinus, supraventricular, ventricular), conduction disturbances, and heart rate variability changes.

Data will be collected on an Excel spreadsheet system. A dedicated hard-copy paper copy of the spreadsheet will be produced and kept as a backup.

Results will be analyzed using the SPSS. A p-value < 0.05 will be considered statistically significant. Descriptive statistical methods will be used to describe key features of groups. Parametric or non-parametric tests (depending on the distribution of the obtained data) will be used for comparing the means and probabilities of two independent populations (Student's t-test, Z-test, or Mann-Whitney U test). When evaluating different diagnostic tests between each other correlation coefficients will be used. Finally, when calculating differences between cardiovascular outcomes/complications - odds ratio assessment (logistic regression, conditional logistic regression) will be done.

Expected outcomes: this study will help evaluate possible long term cardiovascular complications after COVID-19 depending on repolarization changes during the disease and its persistence. These findings could help in the development of long-term monitoring recommendations for patients who have recovered from COVID-19 and forecasting long-term outcomes.

Adverse reactions: The is no expectation of any adverse outcomes or reactions.

Reasons for withdrawal or termination: A subject may be discontinued from the study at any time if the subject feels that it is not in the subject's best interest to continue.

The following is a list of reasons for study discontinuation:

1. Subject withdrawal of consent.
2. Due to temporary or complete withdrawal of researchers or specialists conducting the analysis from the execution of the biomedical study.
3. After collecting the required number of subjects needed to obtain statistically reliable data.
4. If no valuable information is obtained from the primary data.
5. If potential harm to subjects is observed.

All subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice. Reasonable attempts will be made by the Investigators to provide a reason for subject withdrawals.

SAMPLE SIZE JUSTIFICATION Null hypothesis: the frequency of arrhythmias and overall cardiovascular events over two years after the disease in patients who had COVID-19 and changes in ECG ventricular repolarization does not differ from frequency of these events in patients who had COVID-19without changes in ECG ventricular repolarization parameters.

Type I error rate: α=0.05. The required minimum number of subjects to obtain statistically reliable conclusions was calculated using formulas with the 'sample size calculator' (https://sample-size.net/sample-size-means/). The formulas used for comparing means (using the T statistical criterion) and for comparing means of repeated measurements (paired T-test) were applied. A confidence level of 0.95 and a power of 0.8 were chosen for the calculations.

Since participants are planned to be evaluated based on several criteria, the calculations were performed separately for each criterion, and the largest sample size was selected (based on the mean differences in repolarization disorders between those who had and did not have severe COVID-19; the prevalence of repolarization disorders and arrhythmias during the post-recovery period from severe COVID-19. Since this prevalence in the literature ranges from 10% to 27% for this study calculations the investigators chose 15%) Based on the aforementioned criteria, the required sample size of 195 individuals (30 subjects with repolarization disorders and 165 subjects without). was calculated. The number was increased by 10%.

The final number is 215 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient was hospitalized and treated in LUHS Kaunas Hospital for acute COVID-19 2 years ago (starting from 2022 January 1st).
* During hospitalization COVID-19 was verified with PCR test from nasopharyngeal swab.

Exclusion Criteria:

* COVID-19 was not verified with PCR test from nasopharyngeal swab.
* Patients who are unable to give informed consent for participation in study; vulnerable individuals: students if their participation is related to their studies, employees of healthcare institutions subordinate to the researcher, residents of social care institutions, and soldiers during their active military service.
* Patients with an implanted pacemaker or cardioverter-defibrillator.
* Patients whose permanent residence is not in Lithuania and who are not Lithuanian citizens.
* Patients for whom it is not possible to perform ECG and ICG tests due to various circumstances.
* Pregnant individuals (including individuals who were pregnant during the disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will consist of patients who have had COVID-19 and were treated in the LSMU Kaunas Hospital inpatient units two years ago (starting 2024 January 1st). The invitation will be communicated through family doctors to attend a cardiologist's consultation at the LSMU Kaunas Hospital two years after their hospitalization. Those who agree to participate and meet the inclusion criteria and do not have any exclusion criteria will be enrolled. Enrollment will continue until the required sample size is reached.
Sampling Method: Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of arrhythmias (sinus, supraventricular, ventricular) in participants in 2 years after the disease, comparing COVID-19 patients with changes in ECG repolarization parameters and COVID-19 patients without these changes. | In two weeks (14 days) after the enrollment.
  The arrhythmias in medical records and those found during Holter monitoring will be accounted.
  Changes in ECG repolarization parameters are considered present if any of the following are present: prolonged QTc, prolonged Tpec, increased QRS/T angle.
Frequency of ischaemic cardiovascular events in 2 years after the disease, comparing COVID-19 patients with changes in ECG repolarization parameters and COVID-19 patients without these changes. | In two weeks (14 days) after the enrollment.
  The ischaemic events in medical records will be accounted. Changes in ECG repolarization parameters are considered present if any of the following are present: prolonged QTc, prolonged Tpec, increased QRS/T angle.
ECG QTc (measured in milliseconds) during the COVID-19 and after 2 years in individuals who have recovered from COVID-19. | In two weeks (14 days) after the enrollment.
ECG Tpec (measured in milliseconds) during the COVID-19 and after 2 years in individuals who have recovered from COVID-19. | In two weeks (14 days) after the enrollment.
  Tpec = Tpeak-to-Tend interval corrected for heart rate
ECG Tpec/QTc during the COVID-19 and after 2 years in individuals who have recovered from COVID-19. | In two weeks (14 days) after the enrollment.
Changes in ECG QRS-T angle during the COVID-19 and after 2 years in individuals who have recovered from COVID-19. | In two weeks (14 days) after the enrollment.

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: SAP
Time Frame: Starting 6 months after publication